CLINICAL TRIAL: NCT02090621
Title: Extracorporeal Photopheresis After Liver Transplant. Phase II Clinical Trial on Safety and Efficacy in Patients With Progressive Withdrawal of Immunosuppression
Brief Title: Extracorporeal Photopheresis After Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEC-TH; 2012-000633-39 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2014-03-18 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Hepatic Insufficiency
Keywords: Liver; transplantation; Immunosuppression; photopheresis; extracorporeal
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extracorporeal Photopheresis (Experimental): Extracorporeal Photopheresis
  Interventions: Procedure: Extracorporeal photopheresis

INTERVENTIONS:
Procedure: Extracorporeal photopheresis — Extracorporeal photopheresis with Methoxsalen(UVADEX)and immunosuppression reduction Extracorporeal photopheresis (ECP) is an immunomodulatory excellent technical tolerated initially designed for the treatment of cutaneous T-cell lymphoma and various autoimmune diseases, which has been proven effective in reversing episodes acute heart transplants, kidney and lung rejection, and in the treatment of Disease graft versus host both acute and chronic.

SUMMARY:
The purpose of this study is to determine the safety of photopheresis for prophylaxis of allograft rejection in patients who are being withdrawal immunosuppression after liver transplantation.

DETAILED DESCRIPTION:
The photopheresis (ECP) is a therapeutic approach based on the biological effect of ultraviolet light A on mononuclear cells collected by apheresis, and reinfused into the patient.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation 2 years ago
* >18 years
* Treatment with immunosuppression (Cyclosporine or tacrolimus)
* Normal hepatic function during last year
* No acute or chronic rejection
* to have some secondary effect because of immunosuppressors
* Previous disease: alcoholic liver cirrhosis with or without hepatocarcinoma, metabolic disease, amyloid polyneuropathy, hepatitis,cryptogenic cirrhosis and non autoimmune causes
* Signing consent informed form

Exclusion Criteria:

* Additional liver Transplantation
* hypersensitivity to methoxsalen
* Patients with melanoma ,cutaneous carcinoma
* Patients with aphakia
* Patients treated with oxsoralen
* Pregnant women, lactating women or fertile adults that they don´t use a effective anticonception method
* Involved in other assay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events associated with the procedure | 12 months
Non Serious Adverse Events | 12 months
Allograft Rejection | 12 months

SECONDARY OUTCOMES:
Immunosuppressant level | 12 months
  CyA, tacrolimus levels
Liver function test | 12 months
  Total protein, albumin, bilirubin, GOT, GPT, alkaline phosphatase, gamma- GT, Quick index.
Renal Function test | 12 months
  Creatinine, urea, glomerular filtration rate (MDRD), creatinine clearance
Hematological Parameters | 12 months
  Basic hematological parameters:
  Hemoglobin, hematocrit, platelets and leukocytes.
  Metabolic parameters:
  Glucose, uric acid, triglycerides, cholesterol, HDL and LDL cholesterol.
Immunological evaluation | 12 months
  Study of the evolution of subpopulations of blood mononuclear cells peripheral (T cells, B cells and dendritic cells) During removal of the SI measured by flow cytometry of different lymphocyte populations and are expressed as% and / or item # cells / L blood

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Pons, MD, Principal Investigator — Hospital Clínco Universitario Virgen de la Arrixaca
Locations (1):
- Jose Antonio Pons, MD, Murcia, El Palmar, Spain

REFERENCES:
- [Background] Pons JA, Yelamos J, Ramirez P, Oliver-Bonet M, Sanchez A, Rodriguez-Gago M, Navarro J, Bermejo J, Robles R, Parrilla P. Endothelial cell chimerism does not influence allograft tolerance in liver transplant patients after withdrawal of immunosuppression. Transplantation. 2003 Apr 15;75(7):1045-7. doi: 10.1097/01.TP.0000058472.71775.7D. PMID 12698096
- [Background] Pons JA, Ramirez P, Revilla-Nuin B, Pascual D, Baroja-Mazo A, Robles R, Sanchez-Bueno F, Martinez L, Parrilla P. Immunosuppression withdrawal improves long-term metabolic parameters, cardiovascular risk factors and renal function in liver transplant patients. Clin Transplant. 2009 Jun-Jul;23(3):329-36. doi: 10.1111/j.1399-0012.2008.00944.x. Epub 2009 Feb 5. PMID 19210687
- [Background] Pons JA, Revilla-Nuin B, Baroja-Mazo A, Ramirez P, Martinez-Alarcon L, Sanchez-Bueno F, Robles R, Rios A, Aparicio P, Parrilla P. FoxP3 in peripheral blood is associated with operational tolerance in liver transplant patients during immunosuppression withdrawal. Transplantation. 2008 Nov 27;86(10):1370-8. doi: 10.1097/TP.0b013e318188d3e6. PMID 19034005